CLINICAL TRIAL: NCT01558856
Title: Prospective Randomized Trial Comparing Unilateral and Bilateral Neuromodulation Tests in the Treatment of Refractory Idiopathic Overactive Bladder
Brief Title: Unilateral Versus Bilateral Neuromodulation Tests in the Treatment of Refractory Idiopathic Overactive Bladder
Acronym: HAVIR Bi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2011/PW-04; 2012-A00185-38 (Other: ANSM)
Record Dates: First submitted 2012-03-18; First posted 2012-03-20 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2020-08

CONDITIONS: Urinary Bladder, Overactive
Keywords: refractory overactive bladder; neuromodulation; sacral nerves
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unilateral testing (Active Comparator): Following standard procedures, patients in this group will have unilateral testing for neuromodulation of the sacral nerves.
  Intervention: Unilateral electrode placement and testing
  Interventions: Procedure: Unilateral electrode placement and testing
- Bilateral testing (Experimental): Patients in this group will have bilateral testing for neuromodulation of the sacral nerves.
  Intervention: Bilateral electrode placement and testing
  Interventions: Procedure: Bilateral electrode placement and testing

INTERVENTIONS:
Procedure: Unilateral electrode placement and testing — An electrode is placed near a sacral nerve with an anal motor response under general anesthesia. During and adjustment phase, the electode is connected to a test box which allows for adjustment of stimulation parameters. After pinpointing stimulation parameters, the external test box is replaced by an implanted device.
  Arms: Unilateral testing
Procedure: Bilateral electrode placement and testing — Two electrodes are placed, one near each sacral nerve under general anesthesia. During an adjustment phase, the electodes are connected to a test box which allows for adjustment of stimulation parameters. This can result in the use of one or the other, or both electrodes, thus increasing the chances of success and the possibility that the patient is eligible for an implant. After pinpointing stimulation parameters, the external test box is replaced by an implanted device.
  Arms: Bilateral testing

SUMMARY:
The primary objective of this study is to compare the efficacy of unilateral and bilateral neuromodulation tests at 1 month.

DETAILED DESCRIPTION:
The secondary objectives of this study are to compare the following elements between a group of patients undergoing unilater modulation tests (standard procedure) and a group of patients undergoing bilateral neuromodulation tests (experimental procedure) (at 1 month): Pollakiuria, pad use, urge incontinence, symptom severity, % of patients not eligible for an implant, debimetry, tolerance, complications, quality of life.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 1 month of follow-up
* The patient understands and reads French
* The patient has symptoms of overactive bladder resistant to first-line treatments (physiotherapy, anticholinergics)
* The patient suffers from an overactive bladder confirmed by a urodynamic panel
* The patient suffers from an overactive bladder unassociated with bladder obstruction as confirmed by flowmetry
* The patient has primary (idiopathic) overactive bladder primary with normal urinalysis, abdominal and pelvic ultrasound, urine cytology + / - cystoscopy
* The patient has no bleeding disorders, or the disorder is properly controlled after treatment

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* Overactive bladder associated with bladder obstruction as determined by flowmetry
* Overactive bladder unconfirmed by urodynamic panel
* Overactive bladder secondary to another condition:
* vesical: urolithiasis, bladder polyp, interstitial cystitis
* pelivienne: tumor or inflammatory
* neurological: multiple sclerosis, brain tumor, epilepsy
* the patient has an uncorrectable bleeding disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-10-23 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
Success rate | 1 month
  "Success" is defined as a >= 50% improvement in at least one of the following symtoms: pollakiuria, number of urge incontinence episodes with incontinence, number of urge incontinence episodes.

SECONDARY OUTCOMES:
presence/absence: 50% reduction in the number of daily mictions | 1 month
presence/absence: 50% reduction in the number of pads/protections used per day | 1 month
presence/absence: 50% reduction in the number of urge incontinence episodes per day | 1 month
presence/absence: 50% reduction in the number of urge incontinence episodes with incontinence per day | 1 month
Symptom severity as measured by the MHU score | 1 month
  MHU = Mesure Hanicap Urinaire
Yes/no: the patient was eligible for an implant | 1 month
debimetry: flow rate per voiding | 1 month
debimetry: urinary volume per voiding | 1 month
Visual analog scale for pain at the implantation site | 1 month
Visual analog scale for pain due to neuro stimulation (pain in legs or buttocks) | 1 month
Presence/absence of infection of the implant or electrode | 1 month
Change in quality of life: IQoL score | baseline to 1 month
Change in quality of life: KHQ score | baseline to 1 month
Change in quality of life: SF 36 score | baseline to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Wagner, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (6):
- France (6):
  - Clinique Beau Soleil, Montpellier
  - CHU de Nantes - Hôtel Dieu, Nantes
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - APHP - Groupe Hospitalier Pitié-Salpetrière, Paris
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - CHRU de Toulouse - Hôpital de Rangueil, Toulouse

REFERENCES:
- [Result] Wagner L, Alonso S, Le Normand L, Faix A, Kabani S, Castelli C, Game X, Cornu JN, Bey E. Unilateral versus bilateral sacral neuromodulation test in the treatment of refractory idiopathic overactive bladder: A randomized controlled pilot trial. Neurourol Urodyn. 2020 Nov;39(8):2230-2237. doi: 10.1002/nau.24476. Epub 2020 Aug 24. PMID 32835443